CLINICAL TRIAL: NCT00075036
Title: Exploring Patient-Provider Trust Among Individuals With End-Stage Renal Disease
Brief Title: Patient-Provider Trust Among Individuals With End-Stage Kidney Disease
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 040070; 04-CC-0070
Record Dates: First submitted 2003-12-30; First posted 2003-12-31 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09-13

CONDITIONS: Kidney Failure, Chronic
Keywords: Health Disparities; Transplantation; Trust; Interview; Ethnic Bias
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will examine communication and trust between patients in the kidney transplant process and their health care providers. It will assess patients' perception of trust in their physician and nurse coordinator; determine the patients' level of trust in the areas of competence, compassion, control, communication, and confidentiality; and determine how the trust level varies as patients progress in the transplant process.

Patients 18 years of age and older who are in various stages of the kidney transplant process at Walter Reed Army Medical Center and the NIH Clinical Center may be eligible for this study. Candidates include individuals who:

* are on dialysis but not on a transplant waiting list
* are on the organ waiting list and are also on dialysis
* are on the organ waiting list but are not on dialysis
* have had a kidney transplant within the last year.

Participants will be interviewed by someone who is not their direct health care provider about the doctor/patient, primary provider/patient, or nurse/patient relationship, their health history, medical condition, and ideas about their care. With the patient's permission, parts of the interview will be tape-recorded. The interview will take about 30 to 40 minutes.

DETAILED DESCRIPTION:
Health disparities related to the provision of, and access to, healthcare in the United States are well documented across racial and ethnic groups. One area of particular interest to health disparities researchers has been solid organ transplantation. Both provider and patient behaviors are implicated as contributing to ethnic variance of medical care in kidney transplantation. This pilot study will explore the perceptions of trust among patients in the kidney transplant process at the Warren Magnuson Clinical Center at the National Institutes of Health and at Walter Reed Army Medical Center. For sampling purposes the transplant process is defined as 1) patients currently on dialysis; 2) patients on the transplantation waiting list receiving dialysis; 3) patients on the transplantation waiting list not receiving dialysis; 4) patients newly transplanted (less than or equal to one year since transplantation) and 5) patients transplanted for greater than one year. Five dimensions contributing to trust have been identified in the literature: competence, compassion, control, communication and confidentiality. Face-to-face interviews to explore these five dimensions will include questions regarding demographic variables, the Trust in Physician Scale; the Trust in Nurse Scale, and the Patient Trust Scale. Results will be analyzed using descriptive statistics, Chi-square for categorical comparison of means and multivariate analysis for differences between groups.

ELIGIBILITY:
* INCLUSION CRITERIA:

The investigators will interview a cohort of patients from Walter Reed Army Medical Center and the NIDDK intramural program in various stages of the transplant process. The stages are divided into the following categories:

1. individuals on dialysis but not on a waiting list
2. individuals on the organ waiting list who are also on dialysis
3. individuals on the organ waiting list but not on dialysis
4. individuals who have had a kidney transplant within the last year
5. individuals who have had a kidney transplant greater than one year

EXCLUSION CRITERIA:

1. Patients less than 18 years old will not be included in this study. The interview questions and responses to the instruments may be inappropriate for children.
2. All other exclusions are as stated in the NIDDK and WRAMC parent protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2004-02-27; Study Completion 2019-09-13

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Purdie, R.N., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (2):
- United States (2):
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Cain VS, Kington RS. Investigating the role of racial/ethnic bias in health outcomes. Am J Public Health. 2003 Feb;93(2):191-2. doi: 10.2105/ajph.93.2.191. No abstract available. PMID 12554567
- [Background] Furth SL, Garg PP, Neu AM, Hwang W, Fivush BA, Powe NR. Racial differences in access to the kidney transplant waiting list for children and adolescents with end-stage renal disease. Pediatrics. 2000 Oct;106(4):756-61. doi: 10.1542/peds.106.4.756. PMID 11015519
- [Background] Eggers PW. Racial differences in access to kidney transplantation. Health Care Financ Rev. 1995 Winter;17(2):89-103. PMID 10157383